CLINICAL TRIAL: NCT05988970
Title: Impact of Circadian Rhythm on the Spread of Circulating Tumor Cells in Lung Cancer Patients
Acronym: SLEEP_CTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23 POUM 02
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Circadian rhythm; Circulating tumor cells; CTC; CellSearch; ParSortix
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Non- Small Cell Lung Cancer - NSCLC (Other)
  Interventions: Other: Blood samples will be collected at two times before the treatment initiation:

INTERVENTIONS:
Other: Blood samples will be collected at two times before the treatment initiation: — * at 4:00 a.m.
  * at 10:00 a.m.
  Patients will then be followed for data collection for a period of 12 months after inclusion or until disease progression (if applicable).

SUMMARY:
This is a prospective pilot study designed to demonstrate the impact of circadian rhythm on the spread of Circulating Tumor Cells (CTCs) in patients with Non- Small Cell Lung Cancer - NSCLC.

27 patients will be included in the study and will be followed for 12 months.

For each included patient, blood samples will be collected before the anticancer treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed advanced NSCLC (inoperable stage 3 or 4)
2. Patient aged ≥ 18 years
3. Life expectancy > 3 months
4. Patient naïve to treatment for NSCLC
5. Patient hospitalized at least one night for initiation of specific treatment (chemotherapy, radiotherapy, surgery, other...)
6. Patient with no other active cancer. Cancer history accepted if more than 3 years old and considered cured.
7. Patient affiliated to a Social Security scheme in France.
8. Patient having signed informed consent prior to inclusion in the study and prior to any specific study procedure.

Exclusion Criteria:

1. Small-cell cancer or cancer with a majority small-cell contingent
2. Patient previously treated for NSCLC
3. Outpatient
4. Patient with active pathology such as sepsis or uncontrolled inflammatory syndrome
5. Any pathology contraindicating the sample collection procedures required by the study.
6. Pregnant or breast-feeding women.
7. Any psychological, family, geographical or sociological condition that makes it impossible to comply with the medical follow-up and/or procedures stipulated in the study protocol.
8. Patients deprived of their liberty or under legal protection (guardianship, legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
Presence of CTCs detected with the CellSearch technique. | 12 months after the end of inclusions

SECONDARY OUTCOMES:
Quantification of CTCs by the CellSearch technique and expressed in number of cells / millilitre of blood. | 12 months after the end of inclusions
Quantification of CTCs by the ParSortix technique and expressed in number of cells / millilitre of blood. | 12 months after the end of inclusions
Objective response defined as complete or partial response. | 12 months after the end of inclusions
  Response will be assessed according to the clinician's judgment.
Progression-free survival (PFS) defined as the time between the date of inclusion and the date of first progression or death. | 12 months after the end of inclusions

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Larrey, Toulouse
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse